CLINICAL TRIAL: NCT04335422
Title: The Effects of Robot-Assisted Upper Extremity Training on Cognitive and Physical Functions After Stroke: A Randomized Controlled Study
Brief Title: Effects of Robot-Assisted Upper Extremity Training on Cognitive and Physical Functions After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ayşe A Küçükdeveci, MD, Professor of Physşcal Medicine and Rehabilitation, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-313-19
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: stroke; robotic; upper extremity; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective randomized single blind controlled study
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic group (Experimental): Robotic group will receive both routine physical and rehabilitation medicine program and additional upper extremity robot-assisted training by Armeo Spring. Routine physical and rehabilitation medicine program, including physical therapy and exercises, walking and balance training, and occupational therapy to improve activities of daily living will last nearly 2 hours/day and robotic therapy one hour/day. Routine PRM program and robotic therapy will be given through 6 weeks, 5 days a week (A total of 30 sessions of routine PRM program plus robotic therapy).
  Interventions: Device: Robotic group (Upper extremity robot-assisted training plus routine physical and rehabilitation medicine program); Behavioral: Control group (routine physical and rehabilitation medicine program)
- Control group (Active Comparator): Control group will receive only routine physical and rehabilitation medicine program. Routine physical and rehabilitation medicine program, including physical therapy and exercises, walking and balance training, and occupational therapy to improve activities of daily living will last nearly 2 hours/day and will be given through 6 weeks, 5 days a week (A total of 30 sessions of routine PRM program only).
  Interventions: Behavioral: Control group (routine physical and rehabilitation medicine program)

INTERVENTIONS:
Device: Robotic group (Upper extremity robot-assisted training plus routine physical and rehabilitation medicine program) — Upper extremity robot-assisted training will include facilitated shoulder flexion-extension, internal-external rotation, abduction-adduction, elbow flexion-extension, forearm supination-pronation, wrist flexion-extension, ulnar-radial deviation, hand finger flexion-extension movements by means of visual feedback with a 3-dimensional virtual environment in which the patient is asked to perform various tasks such as object reaching, grasping, holding, dropping activities by playing computer games.
  Routine physical and rehabilitation medicine program including physical therapy and exercises, walking and balance training, and occupational therapy to improve daily living activities will be given.
  Arms: Robotic group
Behavioral: Control group (routine physical and rehabilitation medicine program) — Routine physical and rehabilitation medicine program including physical therapy and exercises, walking and balance training, and occupational therapy to improve daily living activities will be given.

SUMMARY:
Stroke is a main cause of disability worldwide. It is characterized by motor and cognitive impairments leading to activity limitations and participation restrictions. Despite improvement in mortality and morbidity following stroke, stroke survivors need access to effective rehabilitation services. Management approach for stroke survivors is classical physical and rehabilitation medicine (PRM) interventions. Nowadays, with the advancement of technology, robotic rehabilitation systems have taken its place among the classical physical and rehabilitation medicine applications. Robotic systems for upper and lower extremity help to improve neuroplasticity by repetitive task-specific activities. Upper extremity robotic systems can be either exoskeleton or end-effector according to their mechanical designs. Exoskeleton robotic systems attach to both proximal and distal segments of the upper extremity (shoulder, elbow, forearm, wrist, fingers) and provide antigravity weight support allowing actuated axes of movements of the upper extremity joints. The system allows the reinforcement and facilitation of movements by means of visual feedback with a 3-dimensional virtual environment in which the patient is asked to perform various tasks by playing computer games. It is reported that robotic therapy can be used complementary to other rehabilitation methods. The neurophysiological effects of robotic therapy were shown to act in the brain, particularly on the primary motor cortex, putamen and capsula interna. The effect on motor recovery was associated with common, synchronous activity involving the corticospinal system. It has been reported by a recent Cochrane review that robot-assisted arm training improves arm function, arm muscle strength and activities of daily living in stroke survivors. A few studies have also reported positive effects on cognitive abilities. However, there are no controlled studies in the literature investigating the effects of robot-assisted upper limb training on cognitive functions following stroke. The aim of this study was to investigate the effects of robot-assisted upper extremity training, applied in addition to the classical PRM program, on cognitive and physical functions after stroke. Primary aim is to investigate the effects on cognitive functions whereas secondary aim is to investigate the effects on upper extremity motor functions and activities of daily living. The investigators hypothesized that adjunctive robotic upper extremity training in addition to classical PRM program would result in better cognitive and physical outcomes compared with the classical PRM program only.

DETAILED DESCRIPTION:
This study is planned as a prospective randomized single blind controlled study. It was approved by the Ethics Committee of Ankara University, Faculty of Medicine and will be conducted in accordance with the Declaration of Helsinki. The study will include 38 stroke survivors who are admitted for rehabilitation at the Department of Physical Medicine and Rehabilitation, Ankara University Medical Faculty. Patients fulfilling the inclusion criteria of the study will randomly be divided into 2 groups as robotic group and control group. Random allocation software (RAS) program will be used to assign the patients to the treatment groups with "block randomization" method and to create the randomization scheme. In this single blinded study, all patients will be evaluated by the same physician (Dr. Merve Dayi). The physician will be blind to patient's assignment. Routine physical and rehabilitation medicine program including physical therapy and exercises, walking and balance training, and occupational therapy to improve activities of daily living will be given to all patients for a total of 6 weeks, 5 days/week, 1 hour/day. Robotic group will additionally receive upper extremity robotic training therapy with Armeo Spring V2.0 exoskeleton (Hocoma Inc.,Zurich, Switzerland) for 6 weeks, 5 days/week, 1 hour/day. The Armeo Spring is an adjustable suspension system for the upper limb that connects to virtual reality, which has settings with several degrees of complexity. The system is an exoskeleton that supports the patient's arm and magnifies any residual active movement of the hemiparetic arm in 3-dimensional space. The patients will receive 30 sessions of robotic therapy under the supervision of physiotherapists, who will adjust the patient's arm and hand in the device and select the virtual reality computer games according to the functional level of the patient's upper limb. All individuals participating in the study will be assessed before and immediately after the treatment and also 3 months at follow-up. Each assessment will include evaluation of cognitive functions, upper extremity motor functions, hand dexterity, upper extremity activities and daily living activities.

Statistical Analysis

As the primary outcome variable, the difference in cognitive functions measured by the Montreal Cognitive Assessment Scale (MoCA) between baseline and post-treatment will be used (Δ MoCA). Group sample sizes of 19 and 19 achieve 80% power to detect a Δ MoCA of 2.4 between robotic and control groups with estimated group standard deviations of 2.5 and 2.5 and with a significance level of 0.05 using a two-sided Mann-Whitney U test. Stratified block randomization will be used to ensure an equal number of subjects in each group. Educational status and age has been chosen as stratification variables. Difference between two groups for continuous variables will be evaluated by Student's t test. Mann-Whitney U test will be used to assess difference between two groups in terms of ordinal variables. The differences in proportions between groups will be compared by using Chi-Square. The repeated-measures ANOVA will be used to test within-group and between-group comparisons for continuous variables and interaction between them. p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients within the age range of 18-80 years
* Patients with subacute stroke (post-stroke duration 1 month - 1 year)
* Patients who have cognitive deficits and who can understand the commands to adapt to robotic training (MMSE ≤ 26)
* Patients with first stroke attack
* Patients who have never received robotic rehabilitation therapy
* Patients with upper extremity (UE) Brunnstrom Stage III and above
* Patients with a spasticity level below 3 (MAS 1-5 assessment system) according to the modified Ashworth Scale (MAS) in the affected upper extremity
* Patients who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

* Patients who cannot understand commands or give informed consent
* Patients without cognitive deficit (MMSE > 26)
* Patients with aphasia
* Patients who do not have sitting balance
* Patients with unilateral neglect
* Patients with unstable systemic medical diseases that may prevent the patient to receive robotic training sessions
* Patients with psychiatric disorders
* Patients with posterior cerebral artery infarction and subarachnoid hemorrhage
* Patients with impaired vision that may affect robotic training
* Patients with a peripheral nerve injury or musculoskeletal disease of the affected upper extremity
* Patients who have pain in the affected upper extremity such that this pain might impede the patient to adapt to robotic training
* Patients with involuntary abnormal movements (e.g. dystonia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Cognitive function | change from baseline at 6 weeks and at 18 weeks
  Cognitive functions will be assessed by "Montreal Cognitive Assessment Scale (MoCA) " which evaluates visuospatial/executive functions, naming, memory, attention, language, abstraction and delayed recall. Total score ranges between 0 and 30. High scores are associated with better clinical outcomes.

SECONDARY OUTCOMES:
Upper extremity motor functions | change from baseline at 6 weeks and at 18 weeks
  "Fugl - Meyer Upper Extremity Motor Rating Scale" will be used to evaluate the motor functions of the upper extremity. It includes 4 subheadings (upper extremity, wrist, hand, coordination/speed). Total score ranges between 0-66 with higher scores predict better outcome.
Hand dexterity | change from baseline at 6 weeks and at 18 weeks
  "Box and Block Test" will be used for assessing manual dexterity. This test is composed of a wooden box divided into two compartments by partition and 150 blocks. The patients are instructed to move as many blocks as possible for a period of 60 seconds. Each hand is scored separately. Higher scores are indicative for better manuel dexterity.
Upper extremity function | change from baseline at 6 weeks and at 18 weeks
  "The Motor Activity Log - 28 (MAG-28)" will be used to asses arm function. This instrument is a structured interview intended to examine how much and how well the subject uses his/her more-affected arm. Total score range between 0-5 and higher scores indicate better function.
Activities of Daily Living | change from baseline at 6 weeks and at 18 weeks
  "Functional Independence Measure (FIM)" will be used to evaluate the functional status of patients in activities of daily living. The FIM's assessment of degree of disability depends on the patient's score in 18 categories, focusing on motor (self care, sphincter control, transfers, locomotion) and cognitive (communication, social cognition) function.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: reference — https://www.ncbi.nlm.nih.gov/pubmed/20400552
- Available data/document: references — https://www.ncbi.nlm.nih.gov/pubmed/28540536